CLINICAL TRIAL: NCT04750681
Title: Evaluation of the Effects of Saffron Extract on Sleep Quality and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comercial Quimica Masso, S.A (Industry)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Saffractiv2019
Record Dates: First submitted 2021-01-28; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Insomnia; Stress
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Each capsule contained 275mg of maltodextrin. Capsules were similar to the saffron investigation product (chlorophyll capsules).
  Interventions: Dietary Supplement: Placebo
- Saffron (Experimental): Each capsule contained 259,5mg of maltodextrin and 15,5mg of saffron extract (Saffr'activ® SAF 3C PIM) that corresponds to 1,6mg of dry saffron extract, 0,9mg of crocins (5.82%) and 0,7mg of safranal (4.6%).
  Interventions: Dietary Supplement: Saffron

INTERVENTIONS:
Dietary Supplement: Placebo — Subjects orally ingested, with water, one capsule per day (in the evening)
  Arms: Control
Dietary Supplement: Saffron — Subjects orally ingested, with water, one capsule per day (in the evening)
  Arms: Saffron

SUMMARY:
Therefore, the aim of this study was to confirm by a randomized double-blind controlled study the beneficial effects of saffron extract (Saffr'activ®) on sleep quality in subjects presenting mild to moderate sleep disorder associated with anxiety.

DETAILED DESCRIPTION:
This study has been designed as a randomized double-blind placebo-controlled interventional study.

Sixty-six subjects were randomly allocated to the control (placebo) or test (Saffr'activ®) group.

A screening visit was scheduled within 4 weeks before Day -7 (study inclusion). At Day -7 and Day 0, questionnaires were completed to evaluate sleep quality, stress level and quality of life. Between Day -7 and Day 0 baseline data for actimeter and sleep diary were registered. Then, subjects were supplemented during 6 weeks with the placebo or saffron (Saffr'activ®) product, depending on their group. Following the baseline period, two other periods of one week were scheduled to collect actigraphy data: between 2 and 3 (from Day 14 to Day 21) weeks and between 5 and 6 (from Day 35 to Day 42) weeks after the beginning of the intervention. At the middle (Day 21) and at the end of the study (Day 42), questionnaires were completed to evaluate sleep quality, stress level and/or quality of life.

ELIGIBILITY:
Inclusion Criteria:

* In good general health as evidenced by medical history and physical examination;
* Presenting mild to moderate chronic primary sleep disorder (evaluated by Insomnia Severity Index - ISI, score between 7 and 21);
* Presenting mild to moderate anxiety (evaluated by Perceived Stress Scale - PSS, score between 6 and 29);
* For women: use of effective contraception;
* Fluent French speaking;
* Provision of signed and dated informed consent form;
* Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Sleep disorders secondary to another health problem;
* Lifestyle habits which would modify the wake-sleep rhythm (e.g. night work) or which would be modified during the study period;
* Pharmacological resistance to common hypnotic drugs or consumption of hypnotic drugs (< 3 months before the inclusion);
* Subjects presenting gastro-intestinal, hepatic, respiratory, psychiatric, kidney or cardiovascular disorders (< 3 months before the inclusion);
* Abnormal blood sampling;
* Subjects presenting depressive disorder (BDI score > 30);
* Recent (< 3 months before the inclusion) change in lifestyle (food, body weight > 5kg, sport);
* Within 3 months before the inclusion, chronic (> 7 days in a row) intake or dosage change of drug(s) or food supplement(s);
* Addict subjects or with historical addiction;
* Subjects who drink more than 3 glasses of alcohol per day (> 30g of alcohol per day);
* Exaggerated consumption of theine (≥ 500ml per day) and caffeine-rich (≥ 400ml per day) beverages and energy drink (≥ 250ml per day);
* Pregnant or lactating woman;
* Known allergy to saffron and/or olives;
* Subjects having participated to another clinical trial one month before the selection visit.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline Leeds Sleep Evaluation Questionnaire score at 42 days | Baseline (day-7 and day 0) and day 42 (end of the study)
  Questionnaire, score 0-100, higher score = better

SECONDARY OUTCOMES:
Change from baseline Leeds Sleep Evaluation Questionnaire score at 21 days | Baseline (day -7 and day 0) and day 21
  Questionnaire, score 0-100, higher score = better
Pittsburgh Sleep Quality Index | Baseline (day -7 and day 0) and day 42 (end of the study)
  Questionnaire, score 0-21, higher score = worse
Epworth Sleepiness Scale | Baseline (day-7 and day 0), day 21 and day 42 (end of the study)
  Questionnaire, score 0-24, higher score = worse
Perceived Stress Scale | Baseline (day -7 and day 0) and day 42 (end of the study)
  Questionnaire, score 0-40, higher score = worse
Short Form (36) Health Survey | Baseline (day -7 and day 0) and day 42 (end of the study)
  Questionnaire, score 0-100, higher score = better
Time in bed | Baseline (from day -7 to day 0), third week (from day 14 to day 21), last week (from day 35 to 42)
  Actimetry
Actual sleep time | Baseline (from day -7 to day 0), third week (from day 14 to day 21), last week (from day 35 to 42)
  Actimetry
Wake after sleep onset | Baseline (from day -7 to day 0), third week (from day 14 to day 21), last week (from day 35 to 42)
  Actimetry
Sleep onset latency | Baseline (from day -7 to day 0), third week (from day 14 to day 21), last week (from day 35 to 42)
  Actimetry
Fragmentation index | Baseline (from day -7 to day 0), third week (from day 14 to day 21), last week (from day 35 to 42)
  Actimetry
Sleep efficiency | Baseline (from day -7 to day 0), third week (from day 14 to day 21), last week (from day 35 to 42)
  Actimetry

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Copine, Dr, Principal Investigator — Université Catholique de Louvain
Locations (1):
- UCLouvain - CICN, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No